CLINICAL TRIAL: NCT04067583
Title: Evaluation of Physician Knowledge of Safety and Safe Use Information for Aflibercept Administered by Intravitreal Injection in Europe: A Follow-up Physician Survey
Brief Title: A Follow-up Physician Survey to Evaluate Physician Knowledge of Safety and Safe Use Information for Aflibercept Administered by Intravitreal Injection in Europe
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20285
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Ophthalmology, Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians with recent aflibercept experience: Ophthalmologists who have prescribed and/or administered aflibercept in the past 6 months
  Interventions: Other: Physician questionnaire

INTERVENTIONS:
Other: Physician questionnaire — This is a one-time cross-sectional survey of physicians, conducted electronically; there are no in person visits

SUMMARY:
With this follow up physician survey researcher want to collect the same data from all participants of the study using a highly structured questionnaire. The questionnaire will gather information related to physician characteristics and experience with Aflibercept, as well as assess physicians' knowledge and understanding of storage and preparation, proper injection technique, and the risks associated with Aflibercept injection into the eye (intravitreal injection). Analysis will be done using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Has signed informed consent
* Is a licensed and practicing ophthalmologist
* Has prescribed and/or administered aflibercept to at least one patient in the past 6 months

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The source of information for the study will be self-reported data collected from physicians using standard questionnaires with closed-ended response choices. Countries included are France, Germany, Italy, Spain, and the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Percentage of physicians responding correctly to each individual knowledge question | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/